CLINICAL TRIAL: NCT04253379
Title: Impact of Executive Functions and Language on Social Cognition in Pediatric Epilepsy
Brief Title: Social Cognition in Pediatric Epilepsy
Acronym: TOMEPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO19122*
Record Dates: First submitted 2020-01-03; First posted 2020-02-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pediatric epilepsy children (Experimental)
  Interventions: Diagnostic Test: Neuropsychological evaluation , Evaluation of theory of mind, Evaluation of executive functions, Evaluation of verbal skills
- healthy children (Active Comparator)
  Interventions: Diagnostic Test: Neuropsychological evaluation , Evaluation of theory of mind, Evaluation of executive functions, Evaluation of verbal skills

INTERVENTIONS:
Diagnostic Test: Neuropsychological evaluation , Evaluation of theory of mind, Evaluation of executive functions, Evaluation of verbal skills — Several tests will be used: Raven's Advanced Progressive Matrices, auditory attention subtest of the NEPSY II, Peabody Picture Vocabulary test, specific comprehension test The cognitive TOM will be evaluated with questions about 4 stories of false beliefs. The affective TOM will be evaluated with a specific emotion inference task 4 adapted subtests from several validated scales will be used to investigate inhibition, cognitive flexibility and working memory The semantic and pragmatic competences will be evaluated with 4 comprehension tasks.

SUMMARY:
The purpose of this study is to investigate the development of social cognition skills in pediatric epilepsy compared to healthy children. There are evidences indicating that children with epilepsy have executive dysfunctions and language problems. Executive functions refer to multiple cognitive processes that contribute to human higher order abilities, such as purposeful and future-orientated behavior. Moreover, the literature regarding development of non epileptic children, with ordinary development indicates that executive functions and language are linked to the emergence of social cognition. Then, the investigators asked if children with epilepsy, as they commonly present executive dysfunctions, would show an atypical development of social cognition. Children with epilepsy and a control group of healthy volunteers will be compared to identify relationships between executive functions, language and social cognition.

DETAILED DESCRIPTION:
Epilepsy is a chronic disorder which affects 50 million people all over the world, with a childhood-onset in 75% of cases. This disorder may interfere with the normal cerebral development and impact cognition skills (Bouis, Cavézian et Chokron, 2011 ; Gallagher et Lassonde, 2005). Executive and language functions are often shown to be affected in previous studies with children with epilepsy (Gencpinar et al., 2015 ; Verrotti, Matricardi, Rinaldi, Prezioso et Coppola, 2015). However, executive functioning and language development are known to be implicated in social cognition acquisitions (Carlson et Moses, 2001 ; Smogorzewska, Szumski et Grygiel, 2018). Yet, less is known about social cognition development in people with epilepsy. Social cognition generally refers to mental operations that underlie social interactions, including perceiving, interpreting, managing, and generating responses to socially relevant stimuli, including the intentions and behaviors others.

The purpose of this protocol is to compare development of social cognition skills, language and executive functions in children with and without epilepsy. This is an observational study; volunteers who participate will not receive any new or experimental therapies. Children in this protocol will undergo an evaluation which may include: a medical history including characteristics of their epilepsy (age at onset, number of antiepileptic drugs, seizure frequency, …) , a nonverbal intellectual efficiency measure , an evaluation of theory of mind, key concept of social cognition, and executive functions then an evaluation of verbal skills .The second purpose of this protocol is to permit the identification of links between development of social cognition and executive et language functions.

Children with epilepsy experience more learning disabilities and behavioral disorders. The treatment of pediatric epilepsy concerns seizure reduction but also reeducation therapy to improve scholar outcome, like speech therapy of psychomotricity. Social consequences may be underestimated in this population, including social cognition.

ELIGIBILITY:
Inclusion Criteria:

* exposed children : children aged 6-12 with a diagnosis of epilepsy French native speaker
* A control group of age-matched children who meet patient selection criteria with the exception of the epilepsy will also be sought

Exclusion Criteria:

* neurological or psychiatric disease in control group
* Raven's Matrices score < percentile 10

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2020-02-02 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
Social cognition evaluation | Day 0
  The cognitive theory of mind test The Cognitive Theory of mind will be evaluated with questions about 4 small stories of false beliefs.
  Number of items : 8 questions Minimum and Maximum values : 0-8 correct responses

SECONDARY OUTCOMES:
Non verbal intellectual efficiency | Day 0
  Raven's Advanced Progressive Matrices It consists of 36 visual geometric designs with a missing piece. In each matrix, the child will select the piece that best completes the pattern.
  Number of items : 36 Minimum and maximum values : 0 - 36 correct responses
Executive functions evaluation | Day 0
  Adaptation of the Flanker Task Executive functions will be evaluated with computized task. For each trial, the child will identify the direction of the central fish. The flanking fish will be pointing in the same direction as the central fish (congruent condition) or in the opposite direction (incongruent condition).
  Number of items : 36 items per condition Minimum and Maximum values : 0 - 1700 millisecondes (Means of Reaction Time)
language evaluation | Day 0
  Peabody Picture Vocabulary Test :
  In each trial, the child will point one picture out of four, the one that best matches a word given by the examiner
  Number of items : 170 Minimum and Maximum values : 0-170 correct responses

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided